CLINICAL TRIAL: NCT05156619
Title: Health Care Disparities in Culturally Diverse, Special Needs & Disadvantaged Populations - Bridging the Gap
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Shani Paluch Shimon, Director, Breast Oncology, Hadassah Medical Organization
Other Study IDs: 060021-HMO-CTIL
Record Dates: First submitted 2021-11-28; First posted 2021-12-14 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Advanced Breast Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Cohort#1: new annual breast cancer cases and cases of recurrence at Hadassah University hospital between 2018-2021 (700)
- Cohort#2: Retrospective study - all clinical trial patients in the Sharett institute of oncology between 1.1.12-30.6.21 (300)
- Cohort#3: all newly diagnosed recurrent/metastatic disease during the study period (200)

SUMMARY:
The overall goal of the project is to characterize the diagnosis, care and outcomes of advanced breast cancer in unique ethnic cohorts in greater Jerusalem, with a focus on the Arab population and ultra-orthodox Jewish population and to improve and streamline care of women from multi-ethnic backgrounds by further understanding barriers to healthcare access. At completion, the collected data will enable planning of culturally appropriate and strategic programs that are culturally tailored to improve the standard of care, outcomes and healthcare access for women living with advanced breast cancer from these unique cohorts.

Target population: Ultra-orthodox Jewish and Arab patients with advanced breast cancer (ABC)

Objectives:

1. Clinical & psychosocial characterization of ultra-orthodox Jewish and Arab women individuals ABC (including clinical characteristic & treatment, outcomes, access and inclusion in clinical trials) along the advanced breast cancer journey
2. Evaluate and identify modes of access to care and barriers to breast cancer care for this population - individually communally, cultural-religiously and professionally (including healthcare professionals)
3. Develop a model for improving health care access and advocacy, tailored to each communities needs
4. Apply the knowledge to developing education training and health promotion - including for the individual, community leadership, and healthcare providers
5. Optimize access to clinical trial participation and reduce any disparities in clinical trial recruitment and participation
6. Develop and tailor culturally appropriate psycho-social interventions to improve psychological wellbeing and quality of life

DETAILED DESCRIPTION:
Project design & methods

The project will include several key aspects with a mixed-methods approach including both qualitative and quantitative data:

Part A - Data Collection

1. A retropective registry of all women with newly diagnosed breast cancer and advanced breast cancer (either de novo or recurrent disease) documenting all clinical disease and treatment characteristics and outcome
2. Gather institutional data on clinical trial recruitment and representation of the ethnic-religious groups under-study. As this is assessed retrospectively, the classification into ethnic-religious sub-groups will be determined by suburb of residence (In Jerusalem ultra-orthodox Jewish and Arab populations in Jerusalem live in distinct homogenous suburbs, distinct from those of the secular Jewish population - this has been demonstrated to be a reliable approach in Jerusalem). Data will be collected on patients recruited between 1/1/2012 until 30/6/2021.
3. Gather data on quality of life, general well-being, spiritual well-being, information receipt along the advanced breast cancer journey for all patients with newly diagnosed advanced breast cancer and compare between the different ethnic groups/cohorts

Part A.1 - Data Collection Methods

1. Data will be collected for a retropective registry of all women with newly diagnosed breast cancer and advanced breast cancer (either de novo or recurrent disease) between 1.1.18-30.6.21 documenting all clinical disease and treatment characteristics and outcome. Data will be collected from the "Mahar" electronic medical record based on lists of all new intakes and all patients with newly recurrent disease that are maintained in the breast oncology unit. Patient identity will be coded and saved anonymously in the data file.

Part A.2 - Data Collection (Appendix 2) Methods Patients documented in the Hadassah "Mahar" to have participated in a clinical oncology trial between 1/1/2012 until 30.6.2021 will be included. Patient identity will be coded and these details will be stored in a separate file. The data collection file will include anonymized patient data. Data collection will include data describing patients' socioeconomic status including gender, date and country of birth, religion, neighborhood and family status. Clinical data about the oncological diagnosis, management and course of disease as well data about the clinical trial intervention and informed consent process will be collected.

Part A.3- Data Collection Quality of Life, Coping and Well-being Method Participants 200 women with metastatic breast cancer will be recruited to the study from Oct 2021 until June 2023. Inclusion criteria: (a) above 18 years old (b) newly diagnosed with metastatic breast cancer or during the last 6 months prior to commencement of the study. Ultra-Orthodox and Arab patients will be part of the study groups, while the secular and national religious patients will serve as control group. Each woman will define her own ethnic/religious identity.

Procedure Patients will be initially approached by the study coordinator during their clinic visit or during their visit to the oncology daycare. They will explained on the study and provide inform consent, which will be storage separately from the study's questionnaires.

Patients who have consented will complete a baseline demographics questionnaire (Appendix 3) and all baseline and ongoing clinical data pertaining to their breast cancer diagnosis and treatment will be collected. Patients will complete psycho-social questionnaires every three months. This will be coordinate by study's coordinator. The questionnaires will be completed using the Qualtrics questionnaire design tool using their personal mobile phone or study's tablet.

Every three months the research coordinator will contact the participant through phone and will either send link to her phone or schedule a meeting in the hospital in which she will answer the questionnaires or answer the questionnaires by phone according to patient's preference.

Some of the Questionnaires will be answered every three months (EORTC QLQ-C30, FACT-B, BDI, FACIT-Sp, STAI) and some will be answered occasionally. The approximate time needed to answer the questionnaire each time will be up to 30 minutes.

The schedule:

Time 1:

* EORTC QLQ-C30
* FACT-B
* BDI
* STAI
* FACIT-Sp
* Demographic questionnaire
* SBI-15R
* ECR-12

Time 2 (month 3):

* EORTC QLQ-C30
* FACT-B
* BDI
* STAI
* FACIT-Sp
* UCLA loneliness scale
* CPASS
* CISC
* Emotional Disclosure and Holding Back subscales
* RAS Time 3(month 6)
* CISC
* Emotional Disclosure and Holding Back subscales
* RAS
* QLQ -INFO25
* Brief Illness Perception Questionnaire
* MAC Time 4(month 9)
* EORTC QLQ-C30
* FACT-B
* BDI
* STAI
* FACIT-Sp
* SCS Time 5 (after month 12)
* EORTC QLQ-C30
* FACT-B
* BDI
* STAI
* FACIT-Sp
* SCS

Questionnaires:

The following questionnaires will be completed every three months:

Quality of Life - The EORTC QLQ-C30 was developed to assess QoL in cancer patients. The 30-item questionnaire includes five functional scales (physical, role, cognitive, emotional, and social), a global quality of life scale, three symptom scales (fatigue, pain, and nausea/vomiting), and several single-item symptom measures (dyspnea, loss of appetite, sleep disturbance, constipation, diarrhea, and financial difficulties). Apart from two items of the global quality of life scale scored on a 7-point scale ranging from 1 (very poor) to 7 (excellent), all items were scored on a 4-point scale ranging from 1 (not at all) to 4 (very much). Higher scores in functioning scales represent a higher level of functioning; higher scores in symptom scales as well as single items, represent a greater level of impairment. Cronbach's α for this instrument was 0.927. There are an official Hebrew and Arabic versions of the questionnaire Well-being - Functional Assessment of Cancer Therapy-Breast (FACT-B) 37-item (Version 4) scale, which contains subscales of physical, social, emotional, and functional well-being in addition to the 10-item breast-specific subscale. The FACT-B total score is the sum of scores of all five subscales. Each item is rated on a 5-point Likert scale. Negatively worded items were recoded such that a higher score indicates as better. There are an official Hebrew and Arabic versions of the questionnaire .

Depression - The Beck Depression Inventory BDI is the most often used self-rating instrument for depressive symptoms. A 21-item self-report depression screening measure. Each item is rated on a 4-point Likert-type scale ranging from 0 to 3, with higher scores indicating higher levels of depression. The measures ask respondents to endorse statements characterizing how they have been feeling throughout the past 2 weeks. The maximum total score for all 21 items is 63. According to the BDI-II manual, scores of 0 to 13 denote minimal depression, scores of 14 to 19 denote mild depression, scores of 20 to 28 denote moderate depression, and scores of 29 to 63 denote severe depression. The questionnaire was found numerous times valid and consistent. There are available Hebrew and Arabic versions of the questionnaire Anxiety - The State-Trait Anxiety Inventory (STAI) is a psychological inventory based on a 4-point Likert scale and consists of 40 questions on a self-report basis. The STAI measures two types of anxiety: state anxiety - anxiety as a response to an event, and trait anxiety - anxiety as a personal characteristic. For the current study we will use only the state subscale. Higher scores represent higher levels of anxiety. The scale was found to have high reliability Spiritual well-being - The FACIT-Sp has three sub-domains of spiritual well-being, which help facilitate an in-depth exploration of the components that constitute spiritual well-being (peace, meaning, and faith). The responses emphasized a sense of meaning in life, harmony, peacefulness, and a sense of strength and comfort from one's faith. It consists of 12 items on 5-point Likert-type scale to measure patient-reported. There are an official Hebrew and Arabic versions of the questionnaire

Demographic and predisposition variables will be measured at Time 1:

Demographic questionnaire was developed for the study and consist of questions regarding socio-demographic variables. It need to be translate into Arabic.

Religiosity - The Systems of Belief Inventory (SBI-15R) was designed to measure religious and spiritual beliefs and practices, and the social support derived from a community sharing those beliefs. The 15-item self-report measure is a revised and shortened form with two dimensions: one with 10 items relating to beliefs and practices, and the second with five items relating to the social support of the religious community. Each item is scored on a four-point scale, ranging from 'strongly disagree' to 'strongly agree'. The score for the total SBI-15 ranges from 0 to 45, with higher numbers indicating more religiosity. Cronbach's alpha is 0.80.

Attachment orientations - participants will complete a shortened version of the Experience in Close Relationships [ECR] Scale. This 12-item version [ECR-12] Likert - scale is based on a previous Hebrew version of the questionnaire and was previously found to be highly reliable. ECR-12 evaluates participants' attachment insecurities through two dimensions: anxiety (e.g. " I need a lot of reassurance that I am loved by people close to me") and avoidance (e.g. "I do not feel comfortable opening to other people") which construct two subscales. A high score on each of the subscales indicates an attachment that is either more anxious or avoidable.

Relational variables will be measured at Time 2. Some of the questionnaire will be answered only by participants that have a spouse.

Loneliness - The revised UCLA loneliness scale is the most widely used instrument to empirically measure the level of loneliness. The UCLA loneliness scale consists 20-item questionnaire that measures loneliness in adults. Each item is rated on a four-point Likert-type scale. Positively worded items are reversed before scoring. Higher scores suggest higher perceived loneliness . Hebrew version is available, but the questionnaire still need to be translated into Arabic.

Perceived social support. The Cancer Perceived Agents of Social Support scale [CPASS; ] was 23 originally developed for Hebrew-speaking participants and consists of 12 items that assess the degree to which a person perceives receiving support from four agents of support: spouse, family, friends, and spiritual community. Three types of support given by each agent of support are assessed, i.e., emotional support, cognitive support, and instrumental support. Answers are given on a 5-point scale, with higher scores indicating higher levels of perceived support. The CPASS has been shown to have adequate validity and reliability.

Questionnaires only for participants that have a spouse:

Contextual self-concealment. Functional Assessment of Cancer Therapy [CISC] consists of 13 items, assessing the frequency of self-concealment behavior in the context of couples coping with a chronic illness. Its wording emphasizes the individual's efforts spent in actively trying to conceal different matters related to the illness (e.g., medical information, physical symptoms, feelings, and implications of the illness), using various methods (e.g., camouflaging illness symptoms, keeping secrets, etc.). Responses are coded on a 7-point scale, ranging from 1 to 7, with higher scores indicating greater frequency of contextual self-concealment. The CISC scale has shown acceptable psychometric qualities. Hebrew version is available, but the questionnaire still need to be translated into Arabic.

Emotional disclosure and holding back of cancer-related concerns. This measure is a modified version of a measure developed by Pistrang and Barker [1995], which was previously used among cancer patients and their spouses. It assesses the degree to which cancer patients and spouses talk to their partners about cancer related feelings and concerns (e.g., "How much did you talk to your spouse/partner about this concern?"). It also assesses the extent to which they hold back from doing so (e.g., "How much did you hold back from talking to your spouse/partner about this concern?"). The questionnaire consists of 10 items, addressing cancer-related concerns (e.g. patient's physical symptoms; cancer treatment; patient's sexual functioning). For each item, respondents will be asked to refer to the past week and rate: a) their level of disclosure, on a 6-point scale and b) their level of holding back, on a 6-point scale. A higher score on the disclosure/holding back subscales indicated a greater level of disclosure/holding back, respectively. This measure has previously demonstrated adequate reliability for both subscales. Hebrew version is available, but the questionnaire still need to be translated into Arabic.

Relationship Assessment Scale (RAS) - The RAS is a short 7-item self-report inventory designed to measure relationship satisfaction. This scale items are rated on a 5-point Likert scale (e.g., "In general, how satisfied are you with your relationship?" and "To what extent has your relationship met your original expectations?"). The RAS is unidimensional and has demonstrated good internal co nsistency. Higher scores represented greater relationship satisfaction. There are available Hebrew and Arabic versions of the questionnaire .

Coping Variables will be measured at Time 3 Information - EORTC Information questionnaire - QLQ -INFO25 QLQ-INFO25 is a 25-item module contains four multi-item scales (information about the disease, medical tests, treatments, and other services) and eight single items (e.g., places of care, self-help to get well, information channels, and information satisfaction and usefulness). QLQ-INFO25 also includes two open questions allowing patients to write about topics of their choice. The response format consisted of a four-point Likert scale (1 - not at all, 2- a little, 3 - quite a bit, 4 - very much), except for the dichotomous (yes/no) questions 51 and 52 and 54 and 55. The questionnaire found to be reliable and valid self-reported instrument. It is used in cross-cultural observational and intervention studies. The questionnaire still needs to be translated into Hebrew and Arabic. The questionnaire will be translated for the current study in forward-backward method.

Illness Perception - Brief Illness Perception Questionnaire consists of nine items, appraising cognitive illness representations, emotional representations and illness comprehensibility. Eight items are rated on Likert scale from 0 to 10. The last item is a causal open-response item, which asks patients to list the three main causal factors in their illness. Responses to the causal item can be grouped into different categories allowing a subsequent categorical analysis. The total score is generated by summing up the scores for the Brief Illness Perception Questionnaire items with a reverse scoring of items 3, 4 and 7. A higher total score reflects a more threatening perception of illness . There are available Hebrew and Arabic versions of the questionnaire Adjustment to Cancer - The Mental Adjustment to Cancer (MAC) Scale is a 40-item self-rating scale on Likert scale of 4 . The scale consists of five subscales: fighting spirit, anxious preoccupation, fatalism, helplessness: hopelessness and avoidance. Previous studies have suggested that the MAC scale has adequate validity and reliability. There are an official Hebrew and Arabic versions of the questionnaire Additional questionnaires will be delivered at Time 4 Self-Compassion- Self-Compassion Scale (SCS) is 25 items and six subscales: Self-Kindness; Self-Judgement; Common Humanity; Isolation; Mindfulness; Over-Identification . Respondents were instructed with the sentence "how I typically act towards myself in difficult times" and are asked to answer each item according to a 5-point scale. Subscale scores are computed by calculating the mean of subscale item responses. Higher scores indicate greater self-compassion. In the original version, the total score showed an excellent internal consistency. There are available Hebrew and Arabic versions of the questionnaire

ELIGIBILITY:
Inclusion Criteria:

* age 18+
* diagnosis of advanced breast cancer within 6 months of study entry

Exclusion Criteria:

* nil

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with with recently diagnosed advanced breast cancer from the greater Jerusalem area treated in Hadassah Medical Centre
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2021-09-26 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Statistical comparisons of all collected demographic and clinical data | 12/2021-6/2023
  Comparative statistical analysis comparing baseline clinical characteristics and survival outcomes between pre-defined socio-ethnic cohorts
Disparities in clinical trial recruitment | 12/2021-6/2023
  comparative analysis of differences in clinical trial recruitment according to pre-defined socio-economic and ethnic background
Temporal changes in quality of life and comparative differences between the pre-defined socio-ethnic groups | 12/2021-6/2023
  Mixed-methods statistical comparison between quality of life changes amongst individuals and between group

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah medical Organization, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No